CLINICAL TRIAL: NCT03104868
Title: Transplant Regimen Adherence for Kidney Recipients by Engaging Information Technologies: The TAKE IT Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Mayo Clinic (Other); Northwestern Memorial Hospital (Other); University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Michael S. Wolf, Associate Division Chief - Division of General Internal Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STU00204465
Record Dates: First submitted 2017-03-28; First posted 2017-04-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplant

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to one of two arms: TAKE IT strategy or usual care.
Who Masked: Participant, Investigator
Masking Description: We will blind: 1) research interviewers involved with outcomes assessment, 2) personnel involved in statistical analyses (Dr. Kwasny, Ms. Patel), 3) principal investigators (Wolf, Ladner). Site project managers will have access to study arm assignments to initiate TAKE IT components to those randomized to receive them.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Patients in this group will receive the usual standard of care.
- Intervention (Experimental): Patients in this group will receive the TAKE IT strategy components.
  Interventions: Behavioral: TAKE IT Strategy

INTERVENTIONS:
Behavioral: TAKE IT Strategy — The TAKE IT Strategy includes:
  1. Programming the electronic health record (EHR) to organize/simplify daily regimen schedules and generate electronic, tangible, print, low literacy medication education materials at every clinical encounter.
  2. SMS text-messaging to remind patients when to take all their medicine.
  3. A web-based patient portal that requests patients to periodically report upon their medication use, providing a continuous link between the transplant center and patient beyond routine in-person visits.
  4. EHR notifications directed to the transplant center nurse coordinator if an adherence-related problem is identified by the web-based portal assessment, who then can activate appropriate staff to respond.
  Arms: Intervention

SUMMARY:
The investigators will evaluate a technology-enabled strategy designed to promote medication adherence, routinely monitor regimen use, and mobilize appropriate transplant center resources to respond early to kidney transplant recipients demonstrating inadequate adherence.

DETAILED DESCRIPTION:
The investigators will evaluate a technology-enabled strategy designed to promote medication adherence, routinely monitor regimen use, and mobilize appropriate transplant center resources to respond early to kidney transplant recipients demonstrating inadequate adherence.

Among patients receiving a kidney transplant (KT), the 5-year risk of organ (graft) failure is high; 30% for deceased donor and 27% for living donor recipients. Medication non-adherence is a leading root cause of graft failure, and KT recipients have the highest reported rate of poor adherence (~35%) among all organ transplant recipients. Despite many attempts, there have been few successful interventions evaluated to date that have significantly improved KT recipients' regimen adherence and subsequent health outcomes over time.

There are many reasons why individuals may not take medication regimens as prescribed, including but not limited to: forgetfulness, misunderstanding, regimen complexity, side effects, health issues, social support, motivation and cost. Therefore no single solution can address all patients. A healthcare team must understand the precise nature of a patient's adherence barriers in order to properly respond. Yet medication adherence is not clinically assessed as part of routine post-transplant care, and prior studies have found that medical staff cannot readily identify poor adherence among patients, let alone the reasons why. Using evidence from the research team's extensive previous studies in other chronic disease contexts, the investigators will implement and comprehensively test a potentially low cost, 'low touch', thus highly scalable intervention: the Transplant regimen Adherence for Kidney recipients by Engaging Information Technologies (TAKE IT) strategy.

The TAKE IT strategy leverages a transplant center's electronic health record and a web-based patient portal, as well as mobile technology to: 1) educate patients on their prescribed Rx regimens, 2) help them organize their daily regimen schedule in the most efficient manner, 3) remind them via Short Message Service (SMS) text when to take their medicine, 4) routinely monitor regimen use, and 5) provide care alerts to engage appropriate transplant center clinical staff (e.g. nurse coordinator, pharmacist, social worker) when medication concerns are detected. All components of the TAKE IT strategy have been developed with prior NIH support, refined with 'user' input (patient, family, clinic staff), and their efficacy tested in non-transplant settings.

The research team's primary aim and hypotheses (H) are to:

Aim 1 Test the effectiveness of the TAKE IT strategy, compared to usual care, to improve KT recipients':

H1 treatment knowledge (indications, potential side effects, demonstrated proper use) H2 medication use (regimen adherence via self-report, pill count, pharmacy records, tacrolimus levels) H3 transplant-specific outcomes (Δ estimated glomerular filtration rate (eGFR), quality of life, re-hospitalization) H4 chronic disease outcomes (blood pressure, HbA1c) They will conduct a 2-arm, patient-randomized controlled trial at two large, diverse transplant centers (Northwestern University; Mayo Clinic). 300 KT recipients within 3 months of transplant ('de novo') and 400 'established' patients between 18 months and 3 years post-KT will be recruited and followed for 2 years (N=700 patients; n=350 per site and n=175 per study arm within each site). In-person interviews will be conducted at baseline, 6, 12, 18 and 24 months. To determine proximal effects of the TAKE IT strategy, a telephone interview will also be administered 6 weeks post-baseline. Electronic health and pharmacy records will be ascertained to capture medication adherence and clinical outcomes.

The secondary aims are to:

Aim 2 Examine the persistence of any effects of the TAKE IT strategy on outcomes over 2 years among new and established KT recipients.

Aim 3 Evaluate the fidelity of each component of the TAKE IT strategy over time, and investigate any patient, provider, or transplant center barriers to implementation.

Aim 4 Determine the costs of delivering the TAKE IT strategy from a transplant center perspective.

Additionally, the investigators will closely evaluate the implementation of all components of the TAKE IT strategy from launch through 2 years follow-up (Aim 2). Their evaluation will include a range of process outcomes to assess the intervention's reliability and sustainability. These findings will determine whether any specific modifications to the TAKE IT strategy are necessary (Aim 3). Finally, the team will estimate the incremental costs of implementing and sustaining the TAKE IT strategy from the perspective of two transplant centers (Aim 4).

ELIGIBILITY:
Inclusion Criteria:

* 1) age 21 or older
* 2) 5 weeks to 24 months post kidney transplant
* 3) English speaking
* 4) primarily responsible for administering own medication
* 5) owns a cell phone and comfortable receiving text messages
* 6) has access to and proficiency using internet in home

Exclusion Criteria:

* any severe, uncorrectable vision, hearing or cognitive impairments

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Mayo Clinic, Arizona, Scottsdale, Arizona
  - Northwestern University, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mellon L, Doyle F, Hickey A, Ward KD, de Freitas DG, McCormick PA, O'Connell O, Conlon P. Interventions for increasing immunosuppressant medication adherence in solid organ transplant recipients. Cochrane Database Syst Rev. 2022 Sep 12;9(9):CD012854. doi: 10.1002/14651858.CD012854.pub2. PMID 36094829
- [Derived] Yoon ES, Hur S, Curtis LM, Wynia AH, Zheng P, Nair SS, Bailey SC, Serper M, Reese PP, Ladner DP, Wolf MS. A Multifaceted Intervention to Improve Medication Adherence in Kidney Transplant Recipients: An Exploratory Analysis of the Fidelity of the TAKE IT Trial. JMIR Form Res. 2022 May 5;6(5):e27277. doi: 10.2196/27277. PMID 35511225

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Patients in this group will receive the Transplant regimen Adherence for Kidney recipients by Engaging Information Technologies (TAKE IT) strategy components.
  TAKE IT Strategy: The TAKE IT Strategy includes:
  1. Programming the electronic health record (EHR) to organize/simplify daily regimen schedules and generate electronic, tangible, print, low literacy medication education materials at every clinical encounter.
  2. Short Message Service (SMS) text-messaging to remind patients when to take all their medicine.
  3. A web-based patient portal that requests patients to periodically report upon their medication use, providing a continuous link between the transplant center and patient beyond routine in-person visits.
  4. EHR notifications directed to the transplant center nurse coordinator if an adherence-related problem is identified by the web-based portal assessment, who then can activate appropriate staff to respond.
Period: Baseline
Arm/Group | Usual Care | Intervention
Started | 225 | 224
Completed | 225 | 224
Not Completed | 0 | 0
Period: 6 Week Follow up
Arm/Group | Usual Care | Intervention
Started | 225 | 224
Completed | 188 | 187
Not Completed | 37 | 37
Not completed — Lost to Follow-up | 5 | 8
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 7 | 6
Not completed — Completed Later Timepoint | 24 | 22
Period: 6 Month Follow up
Arm/Group | Usual Care | Intervention
Started (Participants who started the 6 month period included those who completed the 6 week period and those who were unavailable for the 6 week period.) | 212 | 209
Completed | 188 | 174
Not Completed | 24 | 35
Not completed — Lost to Follow-up | 2 | 2
Not completed — Death | 0 | 1
Not completed — Completed Later Timepoint | 22 | 32
Period: 12 Month Follow up
Arm/Group | Usual Care | Intervention
Started (Participants who started the 12 month period included those who completed the 6 month period and those who were unavailable for the 6 month period) | 210 | 206
Completed | 177 | 171
Not Completed | 33 | 35
Not completed — Lost to Follow-up | 1 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Completed Later Timepoint | 32 | 29
Period: 18 Month Follow up
Arm/Group | Usual Care | Intervention
Started (Participants who started the 18 month period included those who completed the 12 month period and those who were unavailable for the 12 month period) | 209 | 200
Completed | 179 | 165
Not Completed | 30 | 35
Not completed — Lost to Follow-up | 7 | 11
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Graft Loss | 1 | 1
Not completed — Completed Later Timepoint | 19 | 20
Period: 24 Month Follow up
Arm/Group | Usual Care | Intervention
Started (Participants who started the 24 month period included those who completed the 18 month period and those who were unavailable for the 18 month period) | 198 | 185
Completed | 177 | 167
Not Completed | 21 | 18
Not completed — Lost to Follow-up | 15 | 16
Not completed — Death | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Graft Loss | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Patients in this group will receive the TAKE IT strategy components.
  TAKE IT Strategy: The TAKE IT Strategy includes:
  1. Programming the electronic health record (EHR) to organize/simplify daily regimen schedules and generate electronic, tangible, print, low literacy medication education materials at every clinical encounter.
  2. SMS text-messaging to remind patients when to take all their medicine.
  3. A web-based patient portal that requests patients to periodically report upon their medication use, providing a continuous link between the transplant center and patient beyond routine in-person visits.
  4. EHR notifications directed to the transplant center nurse coordinator if an adherence-related problem is identified by the web-based portal assessment, who then can activate appropriate staff to respond.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Intervention | Total
Number analyzed (Participants) | 225 | 224 | 449
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 183 | 186 | 369
  >=65 years | 42 | 38 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (13.3) | 51.7 (12.6) | 51.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 93 | 183
  Male | 135 | 131 | 266
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 44 | 36 | 80
  Not Hispanic or Latino | 177 | 188 | 365
  Unknown or Not Reported | 4 | 0 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 11 | 20 | 31
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 39 | 43 | 82
  White | 161 | 146 | 307
  More than one race | 5 | 9 | 14
  Unknown or Not Reported | 6 | 3 | 9
Recruitment Site [Count of Participants; unit: Participants]
  Northwestern Medicine | 124 | 124 | 248
  Mayo Clinic - Arizona | 101 | 100 | 201
Time Since Transplant [Mean (Standard Deviation); unit: month] | 10.0 (8.2) | 9.7 (8.1) | 9.9 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Rx Pill Count
Description: An in-person pill count using established guidelines will be conducted. When in-person interviews are not possible, pill count will be done over the phone. Adherence will be assessed within drugs. The proportion of pills taken/pills prescribed will be calculated per medication. Patients will be considered non-adherent for a medication if this score is <=80% and adherent if pills taken/pill prescribed>80% (0=non-adherent, 1=adherent).
Time Frame: 1 year - 1.5 years
Population: Analyses included a pill count collected at 1 year or at 1.5 years if a pill count was not collected at 1 year. Observations were excluded if: 1.Medications were not in pill form; 2.Participants couldn't provide accurate quantities on their bottles; 3.Missing Fill or Start Dates, 4.Participants started their medications that day; 5. Pro re nata (PRN) Medications.
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of adherence (1/0)
Units Other Than Participants: Medications
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 178 | 167
Number analyzed (Medications) | 439 | 402
Probability of adherence (1/0) | 0.26 [0.22 to 0.30] | 0.26 [0.22 to 0.30]

2. Secondary Outcome: Correct Medication Dosing Over Past 24 Hours (24 Hour Recall)
Description: Patients are asked to self-report 1) proper dose (# pills), 2) spacing (hours between doses), 3) frequency (times per day), and 4) total pills/day for each prescribed medication over the last 24 hours. Responses are coded as correct or incorrect. Patients will be scored 'yes' if they have demonstrated proper use by correctly reporting all components of the medicine.
Time Frame: 1 year
Population: Observations were excluded if participants did not complete the 24-hour recall questions.
Measure: Least Squares Mean (95% Confidence Interval); unit: Probability of Adherence (1/0)
Units Other Than Participants: Medications
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 166 | 164
Number analyzed (Medications) | 893 | 904
Probability of Adherence (1/0) | 0.89 [0.87 to 0.91] | 0.88 [0.86 to 0.90]

3. Secondary Outcome: Ask-12
Description: The Ask-12 is a self-report scale that assesses general medication attitudes and beliefs. The scale consists of 12 items across three domains (inconvenience/forgetfulness, treatment beliefs, and behaviors), with responses ranging from "Strongly Disagree" to "Strongly Agree". Score can range from 12-60 with higher scores representing greater barriers to adherence.
Time Frame: 1 year
Population: We discovered the wrong timepoint was used in the original analysis. Results were updated in March 2024.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale (12-60)
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 177 | 171
score on a scale (12-60) | 18.4 [17.1 to 19.2] | 17.7 [16.9 to 18.5]

4. Secondary Outcome: Change in Estimated Glomerular Filtration Rate (eGFR), ml/Min/1.73m^2
Description: Change in eGFR (estimated glomerular filtration rate), ml/min/1.73m^2 over 2 years. Values were not adjusted for race.
Time Frame: Value at 2 years minus value at baseline
Population: Participants were analyzed if we were able to retrieve a baseline and 2 year eGFR value from the chart to calculate change. Results were updated in March 2024 after receiving additional data from Mayo Clinic.
Measure: Least Squares Mean (95% Confidence Interval); unit: ml/min/1.73m^2
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 198 | 197
ml/min/1.73m^2 | -0.68 [-2.12 to 0.77] | -0.76 [-2.21 to 0.69]

5. Secondary Outcome: Re-hospitalization
Description: Acute care hospitalizations post transplant. Hospitalizations were self-reported at the 24 month interview and counted if they occurred after the baseline interview.
Time Frame: 2 years
Population: Participants were included if they completed the hospitalization items.
Measure: Least Squares Mean (95% Confidence Interval); unit: probability of re-hospitalization
Arm/Group | Usual Care | Intervention
Number analyzed (Participants) | 173 | 162
probability of re-hospitalization | 0.59 [0.47 to 0.75] | 0.59 [0.46 to 0.75]

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Usual Care | Intervention
All-Cause Mortality (participants affected / at risk) | 6/225 | 6/224
Serious Adverse Events (participants affected / at risk) | 3/225 | 1/224
Other Adverse Events (participants affected / at risk) | 0/225 | 0/224
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=225) | Intervention (N=224)
Graft Loss After Kidney Transplantation (Renal and urinary disorders) | 3 (3) | 1 (1)

LIMITATIONS AND CAVEATS:
Sponsor requested to end enrollment early to focus on retention, with a final sample of 449 participants (700 planned). Therefore were not adequately powered. Due to the Coronavirus disease 2019 (COVID-19) pandemic, in-person interviews became remote resulting in pill count being captured over video or phone instead of an automated pill counter. Many subjects did not bring their medications at baseline as requested, so we were not able to adjust for baseline pill-count adherence as planned.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03104868/Prot_SAP_001.pdf
  • Informed Consent Form (2019-12-10): https://cdn.clinicaltrials.gov/large-docs/68/NCT03104868/ICF_000.pdf